CLINICAL TRIAL: NCT02931448
Title: Occult Carbon Monoxide Poisoning Detection by Pulsated Carboxymetry in an Emergency Department
Acronym: MAS-CO
Status: Withdrawn | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MAS-CO
Record Dates: First submitted 2016-02-19; First posted 2016-10-13 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Carbon Monoxide Poisoning
Keywords: Device assessment
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: Dosage of the blood HbCO thanks to the carboxymeter MASIMO RAD 57

SUMMARY:
In France, the carbon monoxide is one of the first causes of the accidental poisonings with approximately 8000 cases a year, among which 500 deaths.

The severe forms are translated by neurological disorders even a coma or the death straight away. The more insidious forms with a little carboxyhémoglobine level give rise to frustrate clinical pictures, mimicking flu or intestinal syndromes. The syndrome post--intervallaire corresponds to the appearance of remote neuropsychiatric disorders of the poisoning. Its appearance and its gravity are not correlated in the gravity of the initial poisoning, however the precocity of the treatment tends to decrease its frequency.

Carbon monoxide elimination is made under unchanged form in the expired air. In a spontaneous way, the half-life in ambient air is of the order of 4 hours. In ventilation in isobaric pure oxygen, the half-life is shortened at 80 minutes and in hyperbaric oxygen at 23 minutes.

This imposes a fast diagnosis for two reasons:

* For poisonings with low level, the more the investigators wait to measure the carboxyhémoglobine (HBCO), the more they risk not to detect it.
* The oxygen therapy decreases the duration of the poisoning and thus the tissular suffering.

Actually the risk is important to pass next to the diagnosis and to let leave a patient without adapted care and without technical intervention to eliminate the source of the poisoning.

Presently, to make the diagnosis, the investigators possess the analysis of the blood HbCO by realization of gas of the venous blood, which are taken in emergencies, but very often a few hours after the end of the exposure at the source of poisoning, what is translated by a disappearance of the symptoms and an underestimate of the initial blood HbCO. Since 2005, MASIMO laboratory commercialize a pulse carboxymètre, the RAD 57, which allows to estimate the carboxyhémoglobinémie in a not invasive way.

Lot of studies showed the interest of its use in the early screening of carbon monoxide poisonings, allowing a faster dosage of the blood HbCO, and thus an also faster adapted care.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years old consult in ED for :

* cephalalgia
* syncope
* weakness
* nausea
* vomiting
* asthenia

Exclusion Criteria:

* temperature over 38.5 °C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible patients are the ones appearing at emergencies for headaches, nausea and/or vomitings, faintness with or without loss of consciousness, dizzinesses, asthenia, and presenting all the criteria of inclusion and the absence of the criteria of not inclusion.
  Considering the particularity of the foetal poisoning in the carbon monoxide, the pregnant women cannot be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Incidence of poisoning carbon monoxide confirmed | up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers Universitary Hospital, Poitiers, France